CLINICAL TRIAL: NCT02373761
Title: A Prospective Radiostereometric Analysis (RSA) and Clinical Evaluation of the Triathlon Tritanium Total Knee Replacement
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Scott Sporer (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor-Investigator, Scott Sporer, Medical Director, Orthopedic Institute, Central DuPage Hospital
Organization: Central DuPage Hospital (Other)
Other Study IDs: 15-034-CDH
Record Dates: First submitted 2015-02-13; First posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Stryker Triathlon Tritanium primary knee

SUMMARY:
This study seeks to find out if the tibial and patellar components of the Stryker Triathlon Tritanium primary total knee replacement achieve adequate fixation to the underlying bone.

DETAILED DESCRIPTION:
Primary Hypothesis:

The investigators expect the tibial and patellar components of the Stryker Triathlon Tritanium knee to achieve adequate fixation to the underlying bone.

Secondary Hypotheses:

The investigators expect that there will be no continuous migration between one and two years post-operative in the Triathlon Tritanium components.

The investigators expect to see a correlation between radiolucent lines and migration characteristics using RSA.

The investigators expect that inducible displacement exams taken at 2 years post-operative will be able to distinguish between patients identified by RSA measurements as having inadequate fixation.

The investigators expect to see a significant difference in health status and functional outcomes before and after total knee replacement using the Triathlon Tritanium knee.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic osteoarthritis of the knee indicating surgical intervention
* Scheduled to undergo a total knee arthroplasty
* Patients between the ages of 18 and 80, inclusive
* Patient is a candidate for Triathlon Tritanium cementless knee components implanted in accordance with product labeling

Exclusion Criteria:

* Significant co-morbidity affecting ability to ambulate
* Prior arthroplasty, patellectomy or osteotomy with the affected knee
* Active or prior infection of the affected knee
* Morbid obesity (BMI > 40)
* Medical condition precluding major surgery
* Severe osteoporosis
* Neuromuscular impairment
* Pregnancy
* Inability to give informed consent
* Inability to return for follow-up visits for a minimum of two years after surgery
* Currently participating in any other surgical intervention study
* Known allergy to metals
* Flexion contracture greater than 15°
* Extension lag greater than 10°
* Tibial subluxation greater than 10 mm on standing AP radiograph
* Lateral or medial collateral ligament instability (> 10° varus/valgus)
* Leg length discrepancy greater than 10 mm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample of patients undergoing total knee replacement with the Triathlon Tritanium knee components at Central DuPage Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2015-02; Primary Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Radiostereometric analysis of tibial and patellar components of the Stryker Triathlon Tritanium at 6 weeks, 3 months, 6 months, 1 year and 2 years. | 3 years

SECONDARY OUTCOMES:
Improved health status and functional outcomes as measured by the Knee Society Scoring System and EQ-5D questionnaires. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Scott Sporer, MD, Principal Investigator — Central DuPage Hospital
Locations (1):
- Central DuPage Hospital, Winfield, Illinois, United States

REFERENCES:
- [Result] Ryd L, Albrektsson BE, Carlsson L, Dansgard F, Herberts P, Lindstrand A, Regner L, Toksvig-Larsen S. Roentgen stereophotogrammetric analysis as a predictor of mechanical loosening of knee prostheses. J Bone Joint Surg Br. 1995 May;77(3):377-83. PMID 7744919
- [Result] Pijls BG, Valstar ER, Nouta KA, Plevier JW, Fiocco M, Middeldorp S, Nelissen RG. Early migration of tibial components is associated with late revision: a systematic review and meta-analysis of 21,000 knee arthroplasties. Acta Orthop. 2012 Dec;83(6):614-24. doi: 10.3109/17453674.2012.747052. Epub 2012 Nov 9. PMID 23140091